CLINICAL TRIAL: NCT06661135
Title: Total Laparoscopic Versus Open Pancreaticoduodenectomy: a Prospective Comparative Clinical Study
Brief Title: Open Versus Total Laparoscopic Pancreaticoduodenectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Department of general surgery Cairo University (Unknown)
Responsible Party: Principal Investigator, Abdelkarem Ahmed Abdelkarem Mohamed, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pancreaticoduodenectomy
Record Dates: First submitted 2024-10-18; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Pancreatic Neoplasms; Laparoscopic Pancreaticoduodenectomy; Whipple Operation
Keywords: Total laparoscopic pancreaticoduodenectomy; Open vs laparoscopic pancreaticoduodenectomy; Pancreatic neoplasm surgery in developing countries
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: The included patients were equally randomized into two groups: the OPD group, which included patients that would undergo the traditional open procedure, and the LPD group, which included patients that would be subjected to the laparoscopic approach.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator and the outcomes assessor who asses the postoperative pain were not aware of which type of surgery the participant have had.
  Also the pathologist assessing the accuracy of oncology cal resection doesn't know the type of approach that participant had ( open or laparoscopic )
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TLPD (Experimental): This is the group that will receive laparoscopic pancreaicoduodenectomy trocars were inserted (between 5 and 6 trocars were required) and pneumoperitoneum induction was done. The surgeries were performed as previously described . Single loop reconstruction was adopted which involved the formation of all three anastomoses (pancreatico-jejeunostomy, hepatico-jejeunostomy, and gastro-jejeunostomy) on a single jejunal loop. The distance between the hepatico-jejeunostomy, and gastro-jejeunostomy was adjusted at 60 cm for all patients.
  Interventions: Procedure: TLPD total laparoscopic pancreaticoduodenectomy
- OPD (Active Comparator): this group will receive open PD In the OPD group, a bilateral abdominal subcost incision was performed for open surgery
  Interventions: Procedure: OPD open pancreaticoduodenectomy

INTERVENTIONS:
Procedure: TLPD total laparoscopic pancreaticoduodenectomy — It includes removal of the pancreatic or duodenal tumors using the laparoscopy
  Arms: TLPD
Procedure: OPD open pancreaticoduodenectomy — It includes removal of the pancreatic or duodenal tumors using the open technique
  Arms: OPD

SUMMARY:
The goal of this clinical trial is to learn more about Total Laparoscopic pancreaticoduodenectomy ( TLPD ) which is performed for participants with pancreatic tumors using the laparoscope.

TLPD is an operation that includes excision of the tumor with adjacent parts of the head of the pancreas, the duodenum and the part of the external biliary system . In the final step during surgery, and to reconnect the bowel after excision of the tumor, multiple anastomoses or connections will be made by the surgeon.

To get valid results , the investigators performed this randomized controlled trial that compare TLPD with the traditional technique used to remove these tumors through open pancreaticoduodenectomy ( OPD ).

The main questions this study aims to answer are:

Is TLPD superior to open pancraticoduodenectomy ( OPD ) regarding the adequacy of surgical tumor excision ?

Is TLPD lower than OPD regarding the early complications after surgery ?

Researchers will compare participants receiving TLPD with participants receiving OPD regarding :

The time of the operation. The amount of blood lost during surgery. Complications that may happen during or after surgery. Time of recovery after surgery. Duration to amputation. Duration of hospital stay. The adequacy of resection .

DETAILED DESCRIPTION:
Pancreaticoduodenectomy (PD) is a major, complex abdominal surgery that involves removing the pancreatic head together with the common bile duct (CBD) and duodenum. It is usually associated with complications that can severely affect patients' health and lead to mortality.

Pancreaticoduodenectomy is mainly indicated for patients with malignant masses in the head of pancreas and the periampullary region and can be the treatment solution for these patients, providing them with a cure or prolonging their survival. Pancreaticoduodenectomy can also be indicated for some pancreatic cystic neoplasms, particularly intraductal papillary mucinous neoplasms (IPMNs) that can turn malignant, neuroendocrine tumors, metastatic lesions to the pancreas, gastrointestinal stromal tumors, pancreatitis, and major pancreatic injury.

Pancreaticoduodenectomy was not generally accepted until the report introduced by Whipple in 1935 about his successful two-stage PD.. After about five years, Whipple conducted the first anatomic one-stage PD, including an antrectomy and a complete duodenectomy for a pancreatic head tumor.

Pancreaticoduodenectomy has been traditionally performed with an open approach. In 1994, Gagner and Pomp described laparoscopic PD (LPD). In their follow-up study, laparoscopic PD was concluded to have a high conversion rate with no advantages over open PD (OPD). Since then, laparoscopic approaches have been growingly reported, with ongoing research aiming to assess if LPD, being a minimally invasive approach, can improve postoperative morbidity. Nevertheless, LPD is still not broadly accepted. This study aimed to determine the advantages and disadvantages of performing total laparoscopic pancreaticoduodenectomy compared to the open approach.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to the outpatient clinic of Kasr Alainy Hospitals with pancreatic head tumors, duodenal tumors, ampullary, or periampullary tumors who were candidates for either open or laparoscopic pancreaticoduodenectomy
* Patients who accepted to participate in the study.

Exclusion Criteria:

* Patients who were deemed inoperable or irresectable tumors by preoperative investigations.
* Patients with history of previous laparotomies.
* Patients with complex ventral hernias.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | From the date of surgery of every participant to the date of its discharge from hospital or death whichever comes first, assessed up to 3 months .
  Time spent in hospital in days after surgery
Length of postoperative surgical ICU stay | From the date of admission to SICU ( surgical intensive care unit ) after surgery to the date of discharge to ward or death whichever comes first, assessed up to 3 months .
  Length of postoperative surgical ICU stay In days
Amount of blood loss | From start of surgery till skin closure
  Amount of blood lost intraoperative assessed in milliliters
Amount of intraoperative blood transfusion | From start of surgery of every participant till skin closure
  Amount of intraoperative PRBC units transfused intraoperative
30-day mortality | From the date of surgery till one month after
  Reporting Death if happens in the first month postoperatively
Operative time in minutes | From time of skin incision till time of skin closure
  Time spent in surgery

SECONDARY OUTCOMES:
Severity of Postoperative pain | From awakening after surgery ( day 0 ) till ( day 7 ) afterwards
  Assessing postoperative pain daily postoperative using visual analogue score that is a scale of grades from 0 to 10 , with 0 means no pain perceived and 10 indicates the worst pain possible perceived
Gastrointestinal recovery ( time to tolerate oral intake) | From Day two ( D2 ) after surgery for every participant till the date of tolerating oral fluids without vomiting for one complete day , up to two Weeks after surgery
  Time to tolerate oral fluid intake without vomiting . Usually the participants were instructed to take fluids on day 2 after surgery and continue if tolerating and no vomiting occurred for one complete day
Lymph node yield after surgery | It takes 5 days after surgery for the pathological assessment to be completed
  Number of lymph nodes harvested
Ratio of positive lymph nodes to total number of lymph nodes harvested | It takes 5 days after surgery for the pathological assessment to be completed
  Ratio of positive lymph nodes to total number of lymph nodes harvested
State of resection margins after pathological assessment | It takes 5 days after surgery for the pathological assessment to be completed
  State of specimen margins ( free or infiltrated by Tumor )

CONTACTS AND LOCATIONS:
Locations (1):
- Kasralainy school of medicine , Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All scientific individual participant data will be ready for sharing including ( age, sex, associated commorbidies, size of the tumor , time of surgery, type of surgery, hospital stay , SICU stay , resection margin results , units of blood transfusion ,….) abiding in the same time to our local research ethical committee rules
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: For one year starting from the date of acceptance of the paper by a specific , high rank journal
Access Criteria: Any researcher with ORCID number and valid institutional email address
URL: https://mail.google.com/mail/u/0/#inbox

REFERENCES:
- [Derived] Mostafa MS, Hamour D, Aiad GAN, Balamoun HA, Khattab MH, Shazly MN, Nageeb ME, Mohamed AAA. Laparoscopic versus open pancreatoduodenectomy: a pilot randomized trial in a developing African country. Surg Endosc. 2025 Dec 4. doi: 10.1007/s00464-025-12377-x. Online ahead of print. PMID 41345531

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-01): https://cdn.clinicaltrials.gov/large-docs/35/NCT06661135/Prot_SAP_000.pdf